

# TRIAL STATISTICAL ANALYSIS PLAN

Document No.: c42857791-01

BI Trial No.: 1397-0016

Title: A phase I, open-label, single dose, mass balance trial to

investigate metabolism and pharmacokinetics of BI 1291583 (C-14) administered as oral solution in healthy male subjects

Including Protocol Amendment 1 [c37738815-02] Including Protocol Amendment 2 [c37738815-03] Including Protocol Amendment 3 [c37738815-04]

**Investigational** 

BI 1291583

**Product:** 

Responsible trial statistician:

Phone:

Fax:

Date of statistical

20 SEP 2023

analysis plan:

Version: 1.0


Proprietary confidential information

© 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved. This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

# 1. TABLE OF CONTENTS

| TITLE | PAGE | 1 |
|--------------|--------------------------------------------------|----|
| 1. | TABLE OF CONTENTS | 2 |
| LIST O | OF TABLES | 4 |
| 2. | LIST OF ABBREVIATIONS | |
| 3. | INTRODUCTION | |
| 4. | CHANGES IN THE PLANNED ANALYSIS OF THE STUDY | |
| 5.<br>5.1 | ENDPOINTSPRIMARY ENDPOINTS | |
| 5.2 | SECONDARY ENDPOINT | |
| 5.2.1 | Key secondary endpoint | |
| 5.2.2 | Secondary endpoint | |
| 5.3.2 | Safety parameters | 10 |
| <b>6.</b> | GENERAL ANALYSIS DEFINITIONS | |
| 6.1 | TREATMENT | 11 |
| 6.2<br>6.3 | IMPORTANT PROTOCOL DEVIATIONSINTERCURRENT EVENTS | |
| 6.4 | SUBJECT SETS ANALYSED. | |
| 6.6 | HANDLING OF MISSING DATA AND OUTLIERS | |
| <b>6.7</b> | BASELINE, TIME WINDOWS AND CALCULATED VISITS | |
| <b>7.</b> | PLANNED ANALYSIS | |
| 7.1 | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | |
| 7.2<br>7.3 | CONCOMITANT DISEASES AND MEDICATION | |
| 7.3<br>7.4 | TREATMENT COMPLIANCE PRIMARY OBJECTIVE ANALYSIS | 15 |
| <b>7.4.1</b> | Main analysis | |
| 7.5 | SECONDARY OBJECTIVE ANALYSIS | 17 |
| 7.5.1 | Key secondary objective analysis | |
| 7.5.2 | Secondary objective analysis | |
| <b>7.6</b> | FURTHER OBJECTIVE ANALYSIS | |
| 5.63 | | 1= |
| 7.6.2<br>7.7 | Safety parameters EXTENT OF EXPOSURE | |
| I • I | EATENT OF EATOSURE | 1/ |

Date: 20 SEP 2023, Version 1.0

c42857791-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

| 7.8 | SAFETY ANALYSIS | 17 |
|------------|-----------------------------------------------|----|
| 7.8.1 | Adverse Events | |
| 7.8.2 | Laboratory data | |
| 7.8.3 | Vital signs | |
| 7.8.4 | ECG | |
| 7.8.5 | Others | |
| 7.8.5.1 | Physical examination | |
| 7.8.5.2 | Body weight | |
| <b>7.9</b> | OTHER ANALYSIS | |
| 8. | TIMEPOINT OF RELEASE OF TREATMENT INFORMATION | 21 |
| 9. | REFERENCES | 22 |
| 11. | HISTORY TABLE | 24 |

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

# LIST OF TABLES

| Table 6.1: 1 | Analysis phases for statistical analysis of AEs, and actual treatment for | |
|---|---|---|
| | analysis of laboratory data and vital signs | 11 |
| Table 6.4: 1 | Subject sets analysed | 13 |
| Table 11: 1 | History table | 24 |

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

# 2. LIST OF ABBREVIATIONS

| Term | Definition / description |
|---|---|
| AE | Adverse Event |
| AESI | Adverse event of special interest |
| ALT | Alanine aminotransferase |
| AST | Aspartate aminotransferase |
| $AUC_{0	ext{-tz}}$ | Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point |
| BI | Boehringer Ingelheim |
| BMI | Body mass index |
| BP | Blood pressure |
| $C_{max}$ | Maximum measured concentration of the analyte in serum |
| COVID | Coronavirus disease |
| CRF | Case Report Form, paper or electronic (sometimes referred to as 'eCRF') |
| CTP | Clinical trial protocol |
| CTR | Clinical trial report |
| CV | Arithmetic coefficient of variation |
| DILI | Drug induced liver injury |
| ECG | Electrocardiogram |
| EudraCT | European Clinical Trials Database |
| fe <sub>faeces</sub> , 0-tz | Fraction of [14C]-radioactivity excreted in faeces expressed as percentage of the administered dose over the time interval from 0 to the last quantifiable time point |
| fe <sub>urine</sub> , 0-tz | Fraction of [ <sup>14</sup> C]-radioactivity excreted in urine expressed as percentage of the administered dose over the time interval from 0 to the last quantifiable time point |
| gCV | geometric coefficient of variation |
| gMean | Geometric mean |
| ICH | International Conference On Harmonisation |
| IPD | Important protocol deviations |
| LLOQ | Lower limit of quantification |
| MedDRA | Medical Dictionary For Regulatory Activities |


c42857791-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

| Definition / description |
|----------------------------------------|
| Pharmacokinetics |
| Pharmacokinetic parameter analysis set |
| Pulse rate |
| Report appendix generator |
| Residual effect period |
| Report Planning Meeting |
| Serious adverse event |
| Standard Deviation |
| Subject Data Listing |
| System Organ Class |
| Treated set |
| Trial Statistical Analysis Plan |
| Upper limit of normal range |

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

#### 3. INTRODUCTION


As per ICH E9 (1) the purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the revised Clinical Trial Protocol (CTP), and to include detailed procedures for executing the statistical analysis of the primary and secondary variables and other data.

This TSAP assumes familiarity with the CTP and its amendments. In particular, the TSAP is based on the planned analysis specification as written in CTP Section 7 "Statistical Methods and Determination of Sample Size". Therefore, TSAP readers may consult the revised CTP for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size, randomisation.

Study data as collected in the eCRF will be stored in a trial database within the RAVE EDC system. All study data also including external data will then be uploaded to the CDR data warehouse.

| The statistical analyses will be performed within the validated working environmental environment. | onment CARE, |
|---|---|
| including SAS <sup>TM</sup> (current Version 9.4, by | ), and a number |
| of SAS <sup>TM</sup> -based tools (e.g., macros for the analyses of AE data or laboratory | |
| Appendix Generator system (RAGe) for compilation/formatting of the CTR a | appendices). |
| PK parameters will be calculated using Phoenix WinNonlin <sup>TM</sup> software (versor higher, | sion Phoenix 8.1 |

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

# 4. CHANGES IN THE PLANNED ANALYSIS OF THE STUDY

All analyses described in this TSAP are in accordance with the statistical methods described in the revised CTP.

Date: 20 SEP 2023, Version 1.0 BI-VQD-12681 50-415 AD-01 (4.0)

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

#### 5. ENDPOINTS

#### 5.1 PRIMARY ENDPOINTS

Primary endpoints will be the mass balance and total recovery of [<sup>14</sup>C]-radioactivity in urine and faeces, as defined in **Section 2.1.2** of the CTP:

- $fe_{urine,0-tz}$  (fraction of [ $^{14}$ C]-radioactivity excreted in urine expressed as percentage of the administered dose over the time interval from 0 to the last quantifiable time point)
- $fe_{faeces,0-tz}$  (fraction of [ $^{14}$ C]-radioactivity excreted in faeces expressed as percentage of the administered dose over the time interval from 0 to the last quantifiable time point)

Timeframe: The timeframe for determination of these endpoints depends on individual excretion/recovery of radioactivity and may vary between 2 and 6 weeks, inclusive, after drug administration.

#### 5.2 SECONDARY ENDPOINT

### 5.2.1 Key secondary endpoint

Not applicable.


# 5.2.2 Secondary endpoint

The following secondary endpoints will be evaluated for [ $^{14}$ C]-radioactivity, BI 1291583 and five metabolites (M407(1) /BI 1373234, M396(1) / CD 18507, M397(1) / CD 17849, M549(1) / CD 16785) and M141(1) / CD 16426 in plasma, as defined in **Section 2.1.3** of the **CTP**:

- $C_{max}$  (maximum measured concentration of the analyte)
- $AUC_{0-tz}$  (area under the concentration-time curve of the analyte over the time interval from 0 to the last quantifiable time point)



Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.



# **5.3.2** Safety parameters

Safety and tolerability of BI 1291583 will be assessed based on further safety parameters as defined in **Section 2.2.2.2** of the **CTP**:

- Adverse events (including clinically relevant findings from the physical examination)
- Safety laboratory tests
- 12-lead ECG


• Vital signs (blood pressure, pulse rate)



Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

# 6. GENERAL ANALYSIS DEFINITIONS

#### 6.1 TREATMENT


For basic study information on the treatment to be administered, cf. **Section 4** of the **CTP**. Each subject will receive of BI 1291583 (C-14) as an oral solution containing unlabelled BI 1291583 mixed with (C-14) (2% of total dose).



For statistical analysis of AEs, the following analysis phases are defined for each subject.

Table 6.1: 1 Analysis phases for statistical analysis of AEs, and actual treatment for analysis of laboratory data and vital signs

| Study analysis phase | Label | Start (inclusive) | End (exclusive) |
|---|---|---|---|
| Screening <sup>1</sup> | Screening | Date of informed consent | Date/time of administration of study drug |
| On-treatment | BI 1291583 (C-14) | Date/time of administration of study drug | Date/time of administration of study drug + |
| | | | or |
| | | | 12:00 a.m. on day after last contact date (whichever occurs first) |
| Follow up | F/U | Date/time of administration of study drug + | 12:00 a.m. on day after last contact date |

<sup>&</sup>lt;sup>1</sup> See <u>Section 6.7</u> for definition of baseline, which will be used in the statistical analyses of safety laboratory data and vital signs.

AE summary tables will present results for the on-treatment phase only. All AEs will be listed.

Safety laboratory data, vital signs and PK parameters will be analysed with clear differentiation between baseline (cf. Section 6.7) and on-treatment measurements.

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

Measurements will be considered on-treatment, if they were taken within the on-treatment phases as defined in <u>Table 6.1: 1</u>.

More details on the technical implementation of these analyses are provided in the ADS Plan of this TSAP.

#### 6.2 IMPORTANT PROTOCOL DEVIATIONS

Consistency check listings (for identification of deviations from time windows) and a list of protocol deviations (e.g. deviations in drug administration, in blood sampling times, etc.) will be provided to be discussed at the Report Planning Meeting (RPM). At this meeting, it will be decided whether a discrepant data value can be used in analyses, must be corrected in the clinical database or constitutes a PD.

Each protocol deviation must be assessed to determine whether it is an important PD (iPD). For definition of iPDs, and for the process of identification of these, refer to the BI reference document "Identify and Manage Important Protocol Deviations (iPD)" (2) and the DV domain template.

If any iPDs are identified, they are to be summarised into categories and will be captured in the decision log. Categories which are considered to be iPDs in this trial are defined in the DV domain specification. If the data show other iPDs, the definition in the DV domain specification will be supplemented accordingly by the time of the RPM.

IPDs will be summarized and listed. Which kind of iPDs could potentially lead to exclusion from which analysis set is specified in the DV domain specification. The decision on exclusion of participants from analysis sets will be made at the latest at the RPM, after discussion of exceptional cases and implications for analyses. If the data show other iPDs, this table will be supplemented accordingly by the time of the RPM.

Non-important COVID-19 related PDs will only be listed.

A description of handling of iPDs in the analysis is included in the DV domain specification and stored within the TMF in EDMS.

#### 6.3 INTERCURRENT EVENTS

Section is not applicable since no intercurrent events were defined in the CTP.

#### 6.4 SUBJECT SETS ANALYSED


The treated set (TS) and pharmacokinetic parameter analysis set (PKS) will be used as defined in CTP Section 7.2.1.1.

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

Table 6.4: 1 Subject sets analysed

| | Subject | set |
|--------------------------------------|---------|-----|
| Class of endpoint | TS | PKS |
| Disposition | X | |
| iPDs | X | |
| Demographic/baseline characteristics | X | |
| Treatment exposure | X | |
| Primary PK endpoints | | X |
| Secondary PK endpoint | | X |
| Safety parameters | X | |



CTP Section 3.3.4: "If a subject is removed from or withdraws from the trial prior to administration of trial medication, the data of this subject will not be entered in the case report form (CRF) and will not be reported in the clinical trial report (CTR). If a subject is removed from or withdraws from the trial after administration of trial medication, this will be documented and the reason for discontinuation must be recorded in the CRF; in addition, trial data will be included in the CRF and will be reported in the CTR."

**CTP Section 7.3.1**: "It is not planned to impute missing values for safety parameters."

One exception where imputation might be necessary for safety evaluation is AE dates. Missing or incomplete AE dates are imputed according to BI standards ( $\frac{3}{2}$ ).

Missing data and outliers of PK data are handled according to BI standards ( $\frac{4}{2}$ ) and ( $\frac{5}{2}$ ).

**CTP Section 7.3.2**: "PK parameters that cannot be reasonably calculated based on the available drug concentration-time data will not be imputed."

#### 6.7 BASELINE, TIME WINDOWS AND CALCULATED VISITS


In all analyses (safety and PK analyses), the baseline is defined as the last available value prior to study drug administration. Time windows are defined in **Section 6.1** of the **CTP**. Adherence to time windows will be checked at the Report Planning Meeting.


c42857791-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

#### 7. PLANNED ANALYSIS

The format of the listings and tables will follow the BI guideline "Reporting of clinical trials and project summaries" (6).

The individual values of all subjects will be listed. Listings will be sorted by treatment group, subject number and visit (if visit is applicable in the respective listing). AE listings will be sorted by assigned treatment group (see <u>Section 7.8.1</u> below for details). The listings will be contained in Appendix 16.2 (SDL) of the CTR.

The following standard descriptive statistical parameters will be displayed in summary tables of continuous variables:

N number of non-missing observations

Mean arithmetic mean SD standard deviation

Min minimum Median median Max maximum

For plasma and urine concentrations as well as for all PK parameters the following descriptive statistics will additionally be calculated:

CV arithmetic coefficient of variation

gMean geometric mean

gCV geometric coefficient of variation

For PK parameters the following descriptive statistics will additionally be calculated:

P10 10th percentile Q1 1st quartile Q3 3rd quartile P90 90th percentile


The data format for descriptive statistics of plasma and urine concentrations will be identical with the data format of the respective concentrations. The descriptive statistics of PK parameters will be calculated using the individual values with the number of decimal places as provided by the evaluation program. Then the individual values as well as the descriptive statistics will be reported with three significant digits in the CTR.

Tabulations of frequencies for categorical data will include all possible categories and will display the number of observations in a category as well as the percentage (%) relative to the respective treatment group. Percentages will be rounded to integer numbers. The category missing will be displayed only if there are actually missing values. Percentages will be based on all subjects in the respective subject set whether they have non-missing values or not.

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

#### 7.1 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Only descriptive statistics are planned for this section of the CTR. These will be based on the TS.

#### 7.2 CONCOMITANT DISEASES AND MEDICATION

Concomitant diseases and non-drug therapies will be coded according to the most recent version of MedDRA. Concomitant medications and drug therapies will be coded according to the most recent version of the World Health Organisation – Drug Dictionary (WHO-DD). The coding version number will be displayed as a footnote in the respective output.

Only descriptive statistics are planned for this section of the CTR. These will be based on the TS.

**CTP Section 7.2.5:** Previous and concomitant therapies will be presented per treatment group without consideration of time intervals and treatment periods.

A drug or non-drug therapy will be considered concomitant to a treatment, if it

- is ongoing at the time of study drug administration, or
- starts within the analysis phase of the respective treatment (see <u>Section 6.1</u> for a definition of treatments and analysis phases).

The diagnoses and drug as well as non-drug therapies will be listed. Subjects without any concomitant disease or concomitant therapy will be marked with a "No" in the respective column.

The relevance of the concomitant therapies to the evaluation of PK will be decided no later than at the RPM.

#### 7.3 TREATMENT COMPLIANCE

Treatment compliance will not be analysed as a specific endpoint. Any deviations from complete intake will be addressed in the Report Planning Meeting (cf. Section 6.2) and described in the CTR.

**CTP Section 4.3**: "Compliance will be assured by administration of all trial medication in the trial centre under supervision of the investigating physician or a designee. The measured plasma concentrations and/or urinary excretion of trial medication will provide additional confirmation of compliance."

#### 7.4 PRIMARY OBJECTIVE ANALYSIS

#### 7.4.1 Main analysis

The primary and secondary endpoints will be analysed descriptively, as described in the CTP Section 7.2.2 and Section 7.2.3.

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

**CTP Section 7.2.2:** "To avoid underestimation of the total recovery of  $[^{14}C]$ , the excretion during the non-sampling phase of the study will be estimated using linear interpolation between the observed 24-h sampling periods before and after the non-sampling period for urine and faeces respectively."

The analysis of primary and secondary endpoints will be based on the PKS. Subjects in the PKS may not contribute data to every statistical analysis of PK endpoints, in case specific PK endpoints of this subject are missing or excluded for the following reasons.

# Exclusion of PK parameters

The ADS ADPP contains column variables APEX and APEXCO indicating inclusion/exclusion (APEX) of a PK parameter and an analysis flag comment (APEXCO). All analyses based on the PKS are based on PK parameter values which are not flagged for exclusion, i.e. with APEX equal to "Included".

CTP Section 7.2.1.2: "Plasma, urine, faeces, and vomit (as applicable) concentration data and parameters of a subject will be included in the statistical PK analyses if they are not flagged for exclusion due to a protocol deviation relevant to the evaluation of PK (to be decided no later than in the Report Planning Meeting) or due to PK non-evaluability (as revealed during data analysis, based on the criteria specified below). Exclusion of a subject's data will be documented in the CTR."

# Exclusion of PK concentrations


The ADS ADPC (PK concentrations per time-point or per time-interval) contains column variables ACEX or ACEXCO indicating inclusion/exclusion (ACEX) of a concentration and an analysis flag comment (ACEXCO). Exclusion of a concentration depends on the analysis flag comment ACEXCO. For example, if ACEXCO is set to "ALL CALC", the value will be excluded for all types of analyses based on concentrations. If ACEXCO is set to "DESC STATS" the value will be excluded from descriptive evaluations per planned time point/time interval. If ACEXCO contains the addition "TIME VIOLATION" or "TIME DEVIATION", the value can be used for further analyses based on actual times. If ACEXCO is set to "HALF LIFE", the value will be excluded from half-life calculation only; the value is included for all other analyses. Excluded concentration itself will be listed in the CTR associated with an appropriate flag.

Further details are given in "Noncompartmental Pharmacokinetic / Pharmacodynamic Analyses of Clinical Studies" (4) and "Description of Analytical Transfer Files and PK/PD Data Files" (5)



Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.



#### 7.5 SECONDARY OBJECTIVE ANALYSIS

# 7.5.1 Key secondary objective analysis

This section is not applicable as no key secondary objective has been specified in the CTP.

# 7.5.2 Secondary objective analysis

This section is not applicable as no secondary objective has been specified in the CTP.

#### 7.6 FURTHER OBJECTIVE ANALYSIS

#### 7.6.2 Safety parameters

Safety and tolerability will be analysed as described in <u>Section 7.8</u> of this TSAP.

#### 7.7 EXTENT OF EXPOSURE

Since only a single dose is administered per subject, a listing will be sufficient to give account of the extent of exposure.

#### 7.8 SAFETY ANALYSIS

All safety analyses will be performed on the TS.

#### 7.8.1 Adverse Events

AEs will be coded with the most recent version of MedDRA.

The analyses of AEs will be descriptive in nature. All analyses of AEs will be based on the number of subject with AEs and not on the number of AEs.

For further details on summarization of AE data, please refer to "Analysis and Presentation of Adverse Event Data from Clinical Trials" (7) and "Handling of missing and incomplete AE dates" (3).

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

The analysis of AEs will be based on the concept of treatment emergent AEs. That means that all AEs will be assigned to screening, on-treatment or follow-up phases as defined in <u>Section 6.1</u>. AEs will be analysed based on actual treatments on the recorded time of AE onset, as defined in <u>Table 6.1: 1</u>.

An overall summary of AEs will be presented. This summary will include summary statistics for the class of adverse events of special interest (AESIs).

# **CTP Section 5.2.6.1.4**: "The following are considered as AESIs:

# Potential severe DILI

A potential severe Drug Induced Liver Injury (DILI) that requires follow-up is defined by the following alterations of hepatic laboratory parameters:

o An elevation of AST (aspartate aminotransferase) and/or ALT (alanine aminotransferase)  $\geq$ 3-fold ULN combined with an elevation of total bilirubin  $\geq$ 2-fold ULN measured in the same blood sample, or in samples drawn within 30 days of each other, or o Aminotransferase (ALT, and/or AST) elevations  $\geq$ 10-fold ULN

These lab findings constitute a hepatic injury alert and the participants showing these lab abnormalities need to be followed up according to the 'DILI checklist' provided in the ISF. In case of clinical symptoms of hepatic injury (icterus, unexplained encephalopathy, unexplained coagulopathy, right upper quadrant abdominal pain, etc.) without lab results (ALT, AST, total bilirubin) available, the investigator should make sure that these parameters are analysed, if necessary in an unscheduled blood test. Should the results meet the criteria of hepatic injury alert, the procedures described in the DILI checklist should be followed."

The investigator had to classify on the eCRF whether an observed AE was an AESI or not. According to ICH E3 (8), in addition to Deaths, and serious adverse events, 'other significant' AEs need to be listed in the clinical trial report. These will be any non-serious adverse events that led to an action taken with study drug (e.g. discontinuation or dose reduced or interrupted).

The frequency of subjects with AEs will be summarised by treatment, primary SOC and preferred term. Separate tables will be provided for subjects with

- AEs, which were considered by the investigator to be drug related
- SAEs
- AESIs


• AEs summarized by worst intensity.

The SOCs and preferred terms within SOCs will be sorted by descending frequency over all treatment groups.

For disclosure of AE data on ClinicalTrials.gov, the frequency of subjects with non-serious AEs occurring with an incidence of greater than 5 % (in preferred terms) will be summarised

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

by treatment, primary SOC and preferred term. The frequency of subjects with SAEs will also be summarised.

For disclosure of AE data in the EudraCT register, the frequency of AEs, the frequency of non-serious AEs with an incidence of greater than 5 % (in preferred terms) and the frequency of SAEs will be summarized.

For support of lay summaries, the frequency of subjects with drug-related SAEs will be summarized by treatment, primary SOC and preferred term.

# 7.8.2 Laboratory data

The analyses of laboratory data will be descriptive in nature and will be based on BI standards "Handling, Display and Analysis of Laboratory Data" (9).

Analyses will be based on normalised values, which means transforming to a standard unit and a standard reference range. The original values will be analysed if the transformation into standard unit is not possible for a parameter.

Descriptive statistics of laboratory values over time and for the difference from baseline (see <u>Section 6.7</u>) will be provided. Frequency tables of changes between baseline and last value on treatment with respect to the reference range will be presented.

Unscheduled measurements of laboratory data will be assumed to be repeat measurements of the most recent scheduled measurement (e.g. for follow-up or confirmation of a particular value). Therefore, unscheduled measurements will be assigned to the planned time point of the previous scheduled measurement. Descriptive statistics will be calculated by planned time point based on the worst value of the subject at that planned time point (or assigned to that planned time point).

Laboratory data will be compared to their reference ranges. Values outside the reference range will be highlighted in the listings. Possibly clinically significant laboratory values (according to standard BI criteria defining possibly clinically significant abnormalities) will be listed separately.

In general, clinically significant abnormal laboratory values are only those identified either in the Investigator's comments or at the Report Planning Meeting at the latest. With regard to laboratory abnormal values identified at the site it is the Investigator's responsibility to decide whether a lab value is clinically significantly abnormal or not. Those will be reported as baseline conditions (prior to first administration of study treatment) or as AEs (after first administration of study treatment).

#### 7.8.3 Vital signs

The analyses of vital signs (blood pressure and pulse rate) will be descriptive in nature. Descriptive statistics of vital signs over time and for the difference from baseline (see Section 6.7) will be provided.

Date: 20 SEP 2023, Version 1.0 BI-VQD-12681 50-415 AD-01 (4.0)

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

Clinically relevant findings in vital signs data will be reported as baseline conditions (prior to first administration of study treatment) or as AEs (after first administration of study treatment) if judged clinically relevant by the Investigator, and will be analysed as such.

Unscheduled measurements of vital signs will be assigned to planned time points in the same way as described above for laboratory data. However, for vital signs, descriptive statistics will be calculated by planned post-baseline time point based on the last value of the subject at that planned time point (or assigned to that planned time point). If the time of measurement is missing for a scheduled post-baseline measurement (e.g. for follow-up visits) the scheduled measurement will be used in calculation of descriptive statistics (as time difference between scheduled and unscheduled cannot be assessed). If the time of measurement is missing for an unscheduled post-baseline measurement, this measurement will be listed but will be ignored for the calculation of descriptive statistics.

In descriptive statistic of the Screening visit the planned time points will be used. However, if an unscheduled measurement on the same day as the screening visit exists then the unscheduled assessment will be used in descriptive statistics of Screening visit.

#### 7.8.4 ECG

ECG recordings will be checked by the investigator for pathological results. Clinically relevant abnormal findings in ECG will be reported as baseline conditions (at screening) or as AEs (after first administration of study treatment) if judged clinically relevant by the investigator, and will be analysed as such.

No separate listing or analysis of ECG data will be prepared.

#### **7.8.5** Others

# 7.8.5.1 Physical examination

Physical examination findings will be reported as relevant medical history/baseline condition (if a condition already exists before first administration of study treatment) or as AE (if condition emerges after first administration of study treatment) and will be summarized as such.

No separate listing or analysis of physical examination findings will be prepared.

#### 7.8.5.2 Body weight

Body weight will only be listed.

#### 7.9 OTHER ANALYSIS

Not applicable

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

# 8. TIMEPOINT OF RELEASE OF TREATMENT INFORMATION

The treatment information will be loaded into the trial database at trial initiation.

Date: 20 SEP 2023, Version 1.0 BI-VQD-12681 50-415 AD-01 (4.0)

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

# 9. REFERENCES

| 1 | CPMP/ICH/363/96: "Statistical Principles for Clinical Trials", ICH Guideline Topic E9; Note For Guidance on Design, Conduct, Analysis and Evaluation of Clinical Trials, current version |
|---|---|
| 2 | BI-VQD-12045_40-413: "Identify and Manage Important Protocol Deviations (iPD)", current version; KMED |
| 3 | KM Asset BI-KMED-BDS-HTG-0035: "Handling of missing and incomplete AE dates", current version; KMED |
| 4 | KM Asset BI-KMED-TMCP-MAN -0014: "Noncompartmental PK/PD Analyses of Clinical Studies", current version; KMED |
| 5 | KM Asset BI-KMED-TCMP-MAN-0010: "Description of Analytical Transfer Files, PK/PD Data Files and ADA files", current version; KMED |
| 6 | KM Asset BI-KMED-BDS-HTG-0045: "Standards for Reporting of Clinical Trials and Project Summaries", current version; KMED |
| 7 | KM Asset BI-KMED-BDS-HTG-0066: "Analysis and Presentation of Adverse Event Data from Clinical Trials", current version; KMED |
| 8 | CPMP/ICH/137/95: "Structure and Content of Clinical Study Reports", ICH Guideline Topic E3; Note For Guidance on Structure and Content of Clinical Study Reports, current version |
| 9 | KM Asset BI-KMED-BDS-HTG-0042: "Handling, Display and Analysis of Laboratory Data", current version; KMED |

# Boehringer Ingelheim TRIAL STATISTICAL ANALYSIS PLAN 1397-0016


c42857791-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

# 11. HISTORY TABLE

Table 11: 1 History table

| Version | Date<br>(DD-MMM-<br>YY) | Author | Sections changed | Brief description of change |
|---|---|---|---|---|
| 1.0 | 20-Sep-2023 | | None | This is the final TSAP. |